CLINICAL TRIAL: NCT06458335
Title: Addressing Loneliness as a Therapy Target Among Individuals Using Opioids
Brief Title: Intervening on Opioid Use and Loneliness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Medical University of South Carolina (Other); Ohio State University (Other)
Responsible Party: Principal Investigator, Lisham Ashrafioun, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00009396; 1R01DA060966 (NIH)
Record Dates: First submitted 2024-06-09; First posted 2024-06-13 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder; Loneliness; Social Isolation
MeSH Terms: conditions — Opioid-Related Disorders; Social Isolation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive-Behavioral Therapy (Experimental): CBT delivered over the course of 6, ~45 minute sessions delivered via telehealth
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Perceived Social Isolation
- therapist-delivered Health Education (Active Comparator): Health education sessions delivered over the course of 6, ~45 minute sessions delivered via telehealth.
  Interventions: Behavioral: Health Education
- self-guided Health Education (Active Comparator): Health education sessions that are self-guided over the course of 6 sessions
  Interventions: Behavioral: Health Education

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Perceived Social Isolation — 6 sessions focused on addressing thoughts, emotions, and behaviors that maintain feeling alone as a way to reduce loneliness and substance use
  Other Names: CBT-PSI
  Arms: Cognitive-Behavioral Therapy
Behavioral: Health Education — Health education provides information on the importance and benefits of and guidelines for living a health lifestyle
  Arms: self-guided Health Education; therapist-delivered Health Education

SUMMARY:
This study aims to enroll 300 participants who will be assigned to one of three 3 groups. Each group will receive an intervention lasting 6, weekly sessions of 40-60 minutes. Eligibility include having an opioid use disorder and reporting loneliness or feeling alone or disconnected.

DETAILED DESCRIPTION:
Individuals (n = 300) with an opioid use disorder reporting loneliness will be randomized to either (1) therapist-delivered cognitive-behavioral therapy for perceived social isolation, (2) therapist-delivered Health Education, or (3) self-guided Health Education. Loneliness, opioid and other substance use, the amount of social interactions, social support, and mental and physical health factors prior to starting the treatment, after completing the treatment, and 1, 3, and 6 months following the treatment will be assessed to see how well they work compared to each other.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18+
* understand English -have internet access-
* screen positive for an opioid use disorder
* screen positive for elevated loneliness

Exclusion Criteria:

* does not understand consent
* does not have consistent access to a phone and internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in loneliness | Baseline to 6 months
  Loneliness will be measured using the UCLA Loneliness Scale. A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation. Participants rate each item as 1 (never), 2 (rarely), 3 (sometimes) or 4 (often). The scores range from 20-80 with higher scores indicating worse outcome.
Mean change in number of days of opioid use | Baseline to 6 months
  Participants will complete a calendar indicating the type and frequency of drug use.

SECONDARY OUTCOMES:
mean change in social interactions | Baseline to 6 months
  Duke Social Support Index assesses several domains of perceived social support, including social network size, social interaction, social satisfaction, and instrumental social support. Higher scores indicate a higher quality of social interactions. Scores range from 0 to 37.
Mean change in depression | Baseline to 6 months
  Depression will be measured using the PROMIS tool. The scores range from 4-20 with higher scores indicating worse outcome.
Mean change in anxiety | Baseline to 6 months
  Anxiety will be measured using the PROMIS tool. The scores range from 4-20 with higher scores indicating worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data is available upon request through a data use agreement as part of scientific collaboration